CLINICAL TRIAL: NCT03470935
Title: A Non-interventional Study Evaluating the Gynecological Impact of Diagnosis and Treatment of Breast Cancer in Patients Younger Than 40 Years (ARTEMIS)
Brief Title: Non-interventional Study Evaluating Gynecological Impact of Diagnosis and Treatment of Breast Cancer in Patients Younger
Acronym: ARTEMIS
Status: Completed | Type: Observational
Sponsor: Hôpital Privé des Côtes d'Armor (HPCA) (Other)
Responsible Party: Principal Investigator, Jérôme Martin-Babau, Principal Investigator, Hôpital Privé des Côtes d'Armor (HPCA)
Other Study IDs: ARTEMIS
Record Dates: First submitted 2017-10-23; First posted 2018-03-20 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; young women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brest cancer is the most common cancer in women in France with 52.000 new cases diagnosed in 2010 including nearly 6.000 women younger than 40.

The improvement of the fertility conservation of cancer patients is one of the goals put forward by the french Cancer Plan (Objective 8.1).

The issue of fertility after a breast cancer is a frequently raised subjects by the concerned couples today. The improvement in prognosis due to therapeutic advances combined with the increasing age of the first pregnancy and in the recomposed couples bring number of young women between 35 and 40 years followed for breast cancer today to raise these questions with their oncologists.

Young women have a greater risk to develop agressive tumors requiring a mulitimodal treatment whose general and gonadic side effects can be important and permanently impact the reproductive capacity. At the time of diagnosis, almost 50% of these young patients report that they want to consider a later pregnancy but no data are available on the evolution of this wish over time although it is known that anti-cancer treatments have a serious impact on future possibilities of pregnancy(s).

The sequential chemotherapy regimen prescribed in adjuvant or neo-adjuvant situation includes intercaling agents (antracyclines) and an alkylating agent (cyclophosphamide) partially responsible for subsequent fertility disorders. In addition, a chemotherapy-induced amenorrhea (CAI) occurs in 50 to 80% of women according to the studies, the latter is sometines definitive and sequellar of treatment. However, few data describe the time of recovery of menstrual cycles in women with CAI and subsequent impact of fertility.

The aim of this study is to evaluate the impact of cancer diagnosis and treatment on the wishes of fertility before and after the management of cancer of the patients in question, on the recovery of menstrual cycles and the quality of sexual life of these patients.

The investigators hope to improve the pre-therapeutic evaluation of women wishing to implement measures to preserve fertility, to assist women wishing to consider this type of project after cytotoxic treatments and accompany women suffering from a change in self-image that has an impact on their quality of life. These results could help to sensitize the doctors to the difficulties encountered by young women and to improve and/or to strengthen the global and adapted care of these patients.

DETAILED DESCRIPTION:
Selection criteria :

1. Patient with non-metastatic breast cancer ;
2. Age of patient between 18 and 40 years at histological diagnosis ;
3. Patient treated with neoadjuvant or adjuvant chemotherapy with or without radiotherapy or endocrine therapy ;
4. Patient who have completed their chemotherapy and/or radiotherapy treatment for at least 3 months at the time of questionnaire dispatch ;
5. Patient informed of the study (patient must have received the informed consent document and doesn't opposed to it) and who answered to the specific questionnaire of the study ;

Main objective :

=> Describe the impact of diagnosis and the breast cancer care on fertility in patients younger than 40 years.

Secondary objectives :

* Describe the patient population (age, type of histological grade, treatments).
* Describe the recovery of menstrual cycle after chemotherapy (occurrence of menstrual cycles and regularity).
* Describe fertility after treatment.
* Describe the sexual impact (adverse events related to diagnosis and therapeutic care) through an optional part of questionnaire.
* Describe the impact of breast cancer diagnosis on the couple's life.
* Describe the impact on body image (body image satisfaction, breast reconstruction).

ELIGIBILITY:
Inclusion criteria :

1. Patient with non-metastatic breast cancer ;
2. Age of patient between 18 and 40 years at histological diagnosis ;
3. Patient treated with neoadjuvant or adjuvant chemotherapy with or without radiotherapy or endocrine therapy ;
4. Patient who have completed their chemotherapy and/or radiotherapy treatment for at least 3 months at the time of questionnaire dispatch ;
5. Patient informed of the study (patient must have received the informed consent document and doesn't opposed to it) and who answered to the specific questionnaire of the study ;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients aged between 18 and 40 years at the time of diagnosis of non-metastatic breast cancer and having completed their radiotherapy and/or chemotherapy treatment(s) for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Describe the impact of diagnosis and the breast cancer care on fertility in patients younger than 40 years | through study completion, an average of 1 year
  measurement of menstrual cycles

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Martin-Babau, Principal Investigator — Hôpital Privé des Côtes d'Armor (HPCA)
Locations (1):
- Centre investigateur CARIO-HPCA, Plérin, France

IPD SHARING:
Plan to Share IPD: Undecided